CLINICAL TRIAL: NCT01052974
Title: Perioperative Analgesia by Femoral Perineural Catheter for Femoral Neck Fracture - Study KTcol -
Brief Title: Perioperative Analgesia by Femoral Perineural Catheter for Femoral Neck Fracture - Study KTcol
Acronym: KTcol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOI2008-07
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2010-01

CONDITIONS: Femoral Neck Fracture
Keywords: femoral neck fracture; analgesia
MeSH Terms: conditions — Femoral Neck Fractures; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- physiological serum (Placebo Comparator): ropivacaïne controlled by placebo (physiological serum).
  Interventions: Drug: ropivacaine
- ropivacaine (Active Comparator): ropivacaïne controlled by placebo (physiological serum).
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — A widespread collectively practice for the analgesia in prehospital or preoperative period is the single injection of local anesthetic with the technique of the femoral or iliofascial block.
  Intervention: Analgesic treatment using a femoral perineural catheter (inserted from the hospital admission) with continuous infusion of ropivacaïne controlled by placebo.

SUMMARY:
Therapeutic essay of phase IV, monocentric, prospective, randomized, in double-blind during 48 hours(then simple-blind),controlled by placebo.

Abstract:

The increasing incidence of the number of femoral neck fractures and the poor prognosis of this traumatological pathology involves an optimization of the diagnostic, therapeutic and analgesic care.

A widespread collectively practice for the analgesia in prehospital or preoperative period is the single injection ("single shot") of local anesthetic with the technique of the femoral or iliofascial block. Nevertheless the single injection of a dose of local anesthetic associated or not with analgesic adjuvants, due to their pharmacological properties, can't prolong the efficiency of the loco-regional analgesia more than 12 hours.

The aim of our study is to evaluate, in the patients admitted in emergencies for suspicion of femoral neck fractures, the perioperative efficiency of an analgesic treatment using a femoral perineural catheter (inserted from the hospital admission) with continuous infusion of ropivacaïne controlled by placebo (physiological serum).

ELIGIBILITY:
Inclusion Criteria:

* femoral neck fracture

Exclusion Criteria:

* Contraindication with analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03-26 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-11-09 (Actual)

PRIMARY OUTCOMES:
evaluate, in the patients admitted in emergencies for suspicion of femoral neck fractures, the perioperative efficiency of an analgesic treatment using a femoral perineural catheter | from the hospital admission to 24h after surgical operation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BOUHOURS, Principal Investigator — University Hospital, Angers
Locations (1):
- UHAngers, Angers, France

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043